CLINICAL TRIAL: NCT07020572
Title: The iMATTER Project: Preventing Adolescent Depression in Pediatric Primary Care
Brief Title: Improving Mood for Adolescents Through Teaming With End-Users in Routine Care (The iMATTER Project)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: The Klingenstein Third Generation Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-023018
Record Dates: First submitted 2025-06-06; First posted 2025-06-13 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Interpersonal Psychotherapy-Adolescent Skills Training (B-IPT-AST) (Experimental): Brief Interpersonal Psychotherapy-Adolescent Skills Training (B-IPT-AST) is an indicated group depression prevention program adapted from Interpersonal Psychotherapy-Adolescent Skills Training (IPT-AST). In B-IPT-AST, adolescents learn communication (e.g., using I statements, striking while the iron is cold) and interpersonal problem-solving strategies and apply these strategies to their relationships to decrease conflict, increase social support, and improve overall social functioning. B-IPT-AST consists of 1 individual pre-group sessions, 1 individual mid-group session, and 4 group sessions. Parents are invited to attend the mid-group session so the adolescents can apply the interpersonal strategies in a conversation with a parent.
  Interventions: Behavioral: Brief Interpersonal Psychotherapy - Adolescent Skills Training (B-IPT-AST)
- Services as usual (SAU) (Active Comparator): Services as usual (SAU) involves any mental health services adolescents decide to receive in primary care or in the community. It is possible that adolescents in SAU may decide not to participate in any mental health services.
  Interventions: Behavioral: Services as usual (SAU)

INTERVENTIONS:
Behavioral: Brief Interpersonal Psychotherapy - Adolescent Skills Training (B-IPT-AST) — This is an adolescent depression prevention program consisting of 6 sessions (4 group and 2 individual sessions).
  Arms: Brief Interpersonal Psychotherapy-Adolescent Skills Training (B-IPT-AST)
Behavioral: Services as usual (SAU) — Services as usual (SAU) involves any mental health services adolescents decide to receive in primary care or in the community. It is possible that adolescents in SAU may decide not to participate in any mental health services.
  Arms: Services as usual (SAU)

SUMMARY:
This pilot randomized controlled trial will examine the feasibility, acceptability and preliminary efficacy of an adolescent depression prevention program, Brief Interpersonal Psychotherapy-Adolescent Skills Training (B-IPT-AST), in primary care.

DETAILED DESCRIPTION:
Depression is prevalent during adolescence and is associated with negative outcomes. Most adolescent depression prevention programs require significant time and resources. To reduce the research-to-practice gap, the present study will test an adapted version of an evidence-based depression preventive intervention, Interpersonal Psychotherapy-Adolescent Skills Training (IPT-AST), to promote its implementation in primary care (PC). Specifically, a brief, scalable prevention program, Brief IPT-AST (B-IPT-AST), will be tested in a pilot randomized controlled trial in PC. The pilot randomized controlled trial will include adolescents ages 13-17 with subthreshold depression scores on a depression screener, the Patient Health Questionnaire 9-Item: Modified for Teens (PHQ-9-M), completed during an annual PC well-visit. Adolescents will be randomly assigned (2:1 allocation) to B-IPT-AST or services as usual (SAU). Members of the research team will deliver B-IPT-AST. Standardized measures for adolescents and legal guardians will be used to examine emotional outcomes (e.g., depression and anxiety symptoms). Standardized measures will be utilized to assess social processes (e.g., interpersonal conflict). All adolescents randomized to B-IPT-AST will complete a survey measuring acceptability of B-IPT-AST. Additionally, a subset of adolescents who participate in B-IPT-AST will be invited to participate in an hour-long qualitative interview to give feedback on their experiences with B-IPT-AST to inform any further modifications needed to enhance the program's feasibility and acceptability. Feasibility will also be assessed via recruitment and retention information and B-IPT-AST attendance logs.

ELIGIBILITY:
Inclusion Criteria:

For Adolescent Participants

1. Adolescents ages 13 to 17 years.
2. Adolescents must be English-speaking.
3. Legal guardian permission (informed consent) and child consent/assent.
4. A score of 5-10 on the Patient Health Questionnaire 9-Item: Modified for Teens (PHQ-9-M) at the primary care well-visit.
5. Access to a phone, computer, or other electronic device that could be used for study activities

For Legal guardian Participants

1. Legal guardian of an adolescents ages 13 to 17 years who scored 5-10 on the PHQ-9-M at the primary care well-visit.
2. Consent to participate.
3. English-speaking.
4. Access to a phone, computer, and/or tablet to complete remote evaluations.

Exclusion Criteria:

Exclusion criteria will be determined based on electronic health record (EHR) review, eligibility screening questions, the baseline evaluation, and any other interactions with the family.

1. Suicidal ideation or behaviors reported on the PHQ-9-M at their well-visit (score of 1 or higher on item 9 "In the past week, have you had thoughts that you would be better off dead, or of hurting yourself in some way?" and/or yes to either of the supplemental questions which ask, "Has there been a time in the past month when you have had serious thoughts about ending your life?" and "Have you ever, in your whole life, tried to kill yourself or made a suicide attempt?") based on medical record review. For the PHQ-9-M administered at baseline, adolescents who mark yes to the supplemental item about serious suicidal ideation in the past month ("Has there been a time in the past month when you have had serious thoughts about ending your life?") will be excluded.
2. Major medical illness, significant behavioral problems or intellectual or developmental disabilities that may interfere with the completion of all study procedures.
3. Youth may be excluded on a case-by-case basis if the EHR review, eligibility screener, baseline evaluation, or other interactions with the family suggests that the group program would not be appropriate.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Acceptability: A self-report measure, the Attitude Towards Intervention Questionnaire (ATI) | 0-6 Weeks Post-Intervention
  A self-report measure, the Attitude Towards Intervention Questionnaire (ATI), will be completed by adolescents to assess acceptability of Brief Interpersonal Psychotherapy-Adolescent Skills Training (B-IPT-AST) following the intervention. The ATI includes 11 Likert scale items and one open-ended item for providing additional feedback. Likert scales vary by item but are generally 3- or 5-point scales (e.g., very helpful to very unhelpful). Each item is interpreted on its own (e.g., the percentage of teens who found B-IPT-AST very or a little helpful)
Attendance | Weekly during B-IPT-AST
  The number of individual and group B-IPT-AST sessions that teens attend will be tracked in order to report on the average number of group sessions attended (out of 4) for the total sample as well as the average number of individual sessions (out of 2) attended across the sample
Retention | Baseline, 0-6 Weeks Post-Intervention
  To gauge feasibility, retention will be assessed by comparing the number of families who remain in the study through post-intervention to the number who consented.
Depression symptoms | Baseline, 0-6 Weeks Post-Intervention
  Change in depression symptoms will be measured by the Center for Epidemiologic Studies-Depression Scale (CES-D) which assesses the frequency of 20 depressive symptoms over the past week; CES-D scores range from 0 to 60 (scores of 16 or higher are considered elevated); higher scores indicate more depression symptoms
Depression symptoms | Baseline, 0-6 Weeks Post-Intervention
  Change in depression symptoms will also be measured by the Patient Health Questionnaire 9-Item: Modified for Teens (PHQ-9-M). The PHQ-9-M assesses depression symptoms over the past 2 weeks and includes 13 items, 9 of which are included in the total score. Total scores range from 0-27, with higher scores indicating more depression symptoms
Anxiety symptoms | Baseline, 0-6 Weeks Post-Intervention
  Change in anxiety symptoms will be assessed by the Screen for Child Anxiety Related Disorders (SCARED), a 41-item scale assessing symptoms corresponding to different anxiety disorders; the study team will examine total scores and the following subscales: panic, generalized anxiety disorder, and social anxiety; total scores range from 0-82 (25 or higher indicates clinical range); panic scores range from 0-26 (7 or higher indicates clinical range); generalized anxiety disorder scores range from 0-18 (scores of 9 or higher indicates clinical range); social anxiety scale ranges from 0-14 (scores 8 or higher indicate clinical range)

SECONDARY OUTCOMES:
Internalizing and externalizing symptoms | Baseline, 0-6 Weeks Post-Intervention
  Changes in internalizing and externalizing symptoms will be assessed by the Pediatric Symptom Checklist (PSC-17), which will be completed by teens and caregivers; there is a total score (range of 0-34), internalizing subscale (0-24), externalizing subscale (0-20), and attention problems subscale (0-24); higher scores indicate more symptoms
Impairment (Child Report) | Baseline, 0-6 Weeks Post-Intervention
  Change in impairment will be measured via teen report on the Columbia Impairment Scale (CIS), 13-item scale of overall functioning; scores range from 0-52; a score of 15 or higher is considered elevated impairment; higher scores represent greater impairment
Impairment (Parent Report) | Baseline, 0-6 Weeks Post-Intervention
  Change in impairment will be measured via parent report on the Columbia Impairment Scale (CIS), 13-item scale of overall functioning; scores range from 0-52; a score of 15 or higher is considered elevated impairment; higher scores represent greater impairment
Perspective-taking | Baseline, 0-6 Weeks Post-Intervention
  Changes in perspective taking will be measured by the Interpersonal Reactivity Index (IRI), a 7-item perspective-taking scale; scores range from 0-28 with higher scores representing more perspective taking
Social functioning | Baseline, 0-6 Weeks Post-Intervention
  Changes in social functioning will be assessed by the Social Adjustment Scale-Self Report (SAS-SR), a 23-item scale of functioning in school (scores range from 6-30), with friends (scores range from 9-45), with family (scores range from 6-30), and dating (scores range from 2-10); a total score can also be computed (scores range from 23-115); higher scores indicate more difficulties in social functioning
Parent-child conflict (child report) | Baseline, 0-6 Weeks Post-Intervention
  Changes in parent-child conflict will be assessed via teen report on the Conflict Behavior Questionnaire (CBQ), a 20-item questionnaire measuring conflict and negative communication between parents and adolescents; scores range from 0-20; higher scores indicate more conflict
Parent-child conflict (parent report) | Baseline, 0-6 Weeks Post-Intervention
  Changes in parent-child conflict will be assessed via parent report on the Conflict Behavior Questionnaire (CBQ), a 20-item questionnaire measuring conflict and negative communication between parents and adolescents; scores range from 0-20; higher scores indicate more conflict

CONTACTS AND LOCATIONS:
Overall Officials: Molly F Davis, PhD, Principal Investigator — Children's Hospital of Philadelphia, University of Pennsylvania Perelman School of Medicine
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No